CLINICAL TRIAL: NCT06464796
Title: Effectiveness of Motor Imagery Techniques in the Management of Acute Lateral Ankle Sprains in Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01823 Muhammad Ismail Khan
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Ankle Sprains
Keywords: ankle sprains; motor imagery; acute sprians
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Imagery Techniques (Experimental): 1. Motor imagery Techniques
  2. Conventional Therapy
  Interventions: Other: Motor Imagery Techniques
- Conventional Exercise Therapy (Active Comparator): 1. Exercises
  2. Conventional Therapy
  Interventions: Other: Conventional Exercise Therapy

INTERVENTIONS:
Other: Motor Imagery Techniques — * Play a video of person doing a toe-raise exercise where carrying a big barbell on his shoulders.
  * The individual in the video proceeded from a neutral upright position to a tiptoe standing while loud a heavy barbell; the plantar-flexors are used in this workout.
  * The members were said to imagine engaging their ankle flexor muscles in an effort to generate ankle flexion. Both limbs were used during the 10-second imaginary contraction, which was tailed by a 10-second rest. Subsequently five repetitions of the contraction, there was a 30 second pause. Two-minutes of rest were interspersed between five-sets of five-contractions. Fifty imaginary contractions in total.
  Arms: Motor Imagery Techniques
Other: Conventional Exercise Therapy — 1. ROM drills for pronation, flexion and extension.
  2. Ankle strengthening trainings include stand-up on tiptoe, walking on toe-tip, hopping on single foot, and resistance exercise with a latex elastic band.
  3. Proprioceptive exercise include the following exercises: (a) sit on a proprioception board and move the injured limb in a round motion; (b) stand-up with both legs on the board while performing both eyes open and closed; (c) standing with single leg on the board while performing both eyes open; and (d) exercises on a mini-tramp (stand-up on double legs, single leg stances, hops on both left and right legs and on single leg).
  4. Strengthening of the muscles of ankle completed with flexible bands at moderate Intensities.
  5. Training on a stationary bicycle.
  6. lunges forward into a wall.
  7. Steps up and down on the transverse or sagittal plane.
  Arms: Conventional Exercise Therapy

SUMMARY:
To determine the effects of motor imagery techniques on pain, proprioception, instability and strength in acute lateral ankle sprains in soccer players

DETAILED DESCRIPTION:
Football (Soccer) is very a popular game and is played for both leisure and professional occupation. Soccer that is one of the contact game and the main portion of the players life is mostly spend on the sport ground in circumstances where there is a great risk of physical injury. Soccer player requires to be fit physically and mentally in order to cater the outstanding demands of game and training which includes the exceptional levels of attention, memory, and planning, and other diverse mental roles though good proprioception is a vital prerequisite for a good game performance and locomotor system injuries and mild traumatic brain injury. The ankle is contemplated majorly susceptible joint to injure throughout games. About 30% of games injuries including running, contact, and jumping are ankle injuries, and ankle ligamentous injuries account for 77% of ankle injuries. Repetitive occurrence of ankle ligamentous injuries cause prolong injury in the sensory-motor function and proprioceptive, by creating a deficit in the Neuro-muscular reflex response time. In 20% of the cases, repeated ankle ligamentous events can result in unstableness of the ankle joints.

Motor imagery is an active procedure during which the representation of an exact action is internally reproduced within the working memory, deprived of any motor output. Evidence has been presented by Functional imaging studies that during motor imagery like anatomical substrates get activated as during motor performance and exercise, motor imagery has been indicated to boost motor performance and muscle potential. Imagery has also been mentioned to be an effectual adjunctive procedure to physiotherapy programs. The imagery program is utilized to assist members to control, see, and vividly construct an image with in the mind. Motor imagery method form a nerve network, hence motor images boost dynamic balancing capability by facilitation the coordination, proprioceptive sense, and kinesthesia capability. Besides, other researchers have described reduction in pain when imagery has been implemented to other medical disorders.

A study reported that a therapy plus imagery group had better functional retrieved than a control therapy group, during imagery there are extensive activation of neural and muscular mechanisms as if the arm were actually being utilized. Motor imagery was effectual by indicating slow down onset time of peroneal muscle in patients with functional ankle unstableness. MI may be effective for pain relief and development in range of motion among prolong musculoskeletal discomfort condition. MI protocol can be helpful to rehabilitation plans after total knee arthroplasty, as it mainly aids to reduce uneasiness and increase strength. For patients who have had arthroplasty, this pilot study advises that MI therapy should be comprised to the orthopedic treatment. We observed at a few developments brought about by MI on motor retrieval following peripheral injury, mostly in the initial postop phase. Plantar-flexor muscles' voluntary torque cohort was importantly increased by MI training of lower limb muscles, and this force surge was not the result of general motivational effects. When it comes to the rehabilitation of grade II ankle ligamentous tears, MI might be useful.

The management of MSK pain situations has seen a rise in the application of MI in modern years. This study aimed to relating the consequence of motor imagery as an adjunct to standard rehab (intervention) and with standard rehab only (comparison) on ankle pain, instability, strength, proprioception (outcomes) in soccer player with acute lateral ankle sprain (participants). This will help set the foundation for further study and designing treatment protocols of the said population.

ELIGIBILITY:
Inclusion Criteria:

* Active Male football player.
* Age among 18-30 years.
* Football players who had recent lateral ankle sprain allocation accomplished within 72 hours after the sprain.
* Participant had at least one of these symptoms: pain, inflammation, contusion or unable to perform physical activities for more than a day.
* Football players with a history of acute ankle sprains and a self-declared feeling of instability with a Cumberland ankle instability tool score of <27.
* Players who were referred by Rheumatologist/Sports Physiatrist.

Exclusion Criteria:

* Ankle sprain related with lower extremity fracture.
* Other lower extremity injuries.
* Neurological/ Claudication or vascular abnormalities

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 3 weeks
  A Visual Analogue Scale (VAS) is an instrument which evaluates that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured
Cumberland Ankle Instability Test questionnaire | 3 weeks
  Cumberland Ankle Instability Test questionnaire (CAIT) is a 9-items and 30-points scale, to determine the FAI severity
Star Excursion Proprioception Test | 3 weeks
  The SEBT is a valid test that needs participants with maximum strength, Plibility, and proprioception. The objective is to sustain stance on single leg while reaching as far as possible with the opposite leg
Manual Muscle Testing | 3 weeks
  Muscle testing is an important examination tool to assess diminishment and shortfall in muscle performance, including strength, power, or endurance

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmed Awan, PhD, Study Chair — Riphah International University
Locations (1):
- Hayatabad Sports Complex, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No